CLINICAL TRIAL: NCT06224998
Title: Comparison of the Effects of Schroth and Pilates Exercises on Respiratory Functions, Functional Capacity, Balance, Spine Structure and Quality of Life in Idiopathic Adolescent Scoliosis
Brief Title: Schroth and Pilates Exercises in Idiopathic Adolescent Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, kevser kacmaz, research asisstant, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: scoIzmirKCU
Record Dates: First submitted 2023-12-11; First posted 2024-01-25 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Schroth exercises (Experimental): Schroth technique, one of these exercise approaches, is primarily based on isometric muscle contraction exercises that aim to rotate, lengthen and stabilize the spine. The key component of the Schroth method is autocorrection, defined as the patient's ability to reduce spinal deformity through active postural realignment of the spine in three dimensions. Automatic correction is achieved through self-extension and specific segmental corrections adapted to each curve pattern. The International Scoliosis Orthopedic Treatment and Rehabilitation Association considers automatic correction to be the most important element of scoliosis-specific exercise therapy.
  Interventions: Behavioral: Exercise
- Pilates exercises (Experimental): Pilates exercise training improves flexibility and overall physical health by emphasizing strength, posture and coordination of respiratory-related movements. Pilates improves body awareness by working the body as a whole, using gravity and springs to increase resistance and assist in the execution of movements. Pilates, used in neuromuscular training and functional activity training in physiotherapy, is widely used for stimulation of blood circulation, development of flexibility, muscle endurance and strength, postural harmony and body awareness. Pilates has been reported to be an effective physical technique for pain, symptom management, and improving the Cobb angle in scoliosis. Pilates has been reported to be effective in improving scoliosis by correcting poor posture, strengthening the muscles necessary for postural correction, and maintaining body balance.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise is the most appropriate treatment for low and moderate AIS cases due to its low cost and low risk of complications. Exercises prevent the development of many problems by controlling the severity of curvature and preventing the progression of curvature. It is thought that scoliosis exercises can delay or even prevent surgery and reduce the duration or degree of brace, especially in patients with low-to-moderate curvature during growth. One of these exercise approaches, the Schroth technique, is primarily based on isometric muscle contraction exercises that aim to rotate, lengthen and stabilize the spine. The core component of the Schroth method is autocorrection, defined as the patient's ability to reduce spinal deformity through active postural realignment of the spine in three dimensions.

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a common anomaly that is frequently seen in prepubertal growth and is characterized by deviation and rotation of the spine, causing high level of disability. Pubertal development and asymmetrical load distribution increase the progression of the deformity. Affecting the spinal structure and its movement can affect the structures and cause problems in many areas such as pain, balance, respiration, mental health and quality of life. AIS can cause functional disability by causing deterioration in chest wall mechanics, weakness in respiratory muscles and limitation of functional capacity. As the disease progresses, prolonged hypoinflation and atelectasis lead to irreversible atrophy of the lungs and further reduction in lung volume. Displacement and/or compression of the heart due to thoracic deformity may not allow for the required increase in stroke volume during exercise. In severe cases, patients are at risk of developing pulmonary hypertension due to chronic respiratory failure and chronic atelectasis, chronic hypoxemia, chronic hypercapnia. In addition, muscle atrophy and muscle weakness in AIS are thought to cause muscle imbalances and loss of balance.

Exercise is the most appropriate treatment for low and moderate AIS cases due to its low cost and low risk of complications. Exercises prevent the development of many problems by controlling the severity of curvature and preventing the progression of curvature. It is thought that scoliosis exercises

can delay or even prevent surgery and reduce the duration or degree of brace, especially in patients with low-to-moderate curvature during growth. One of these exercise approaches, the Schroth technique, is primarily based on isometric muscle contraction exercises that aim to rotate, lengthen and stabilize the spine. The core component of the Schroth method is autocorrection, defined as the patient's ability to reduce spinal deformity through active postural realignment of the spine in three dimensions.

Another frequently used exercise method, Pilates exercise training improves flexibility and overall physical health by emphasizing the coordination of movements associated with strength, posture, and breathing. However, the effects of these exercises in reducing curvature and related problems are controversial in the literature. Therefore, in this study, we aimed to investigate the effects of Schroth and pilates exercises on respiratory functions, functional capacity, balance, spine structure and quality of life in adolescents with idiopathic scoliosis.

Thirty patients aged 10 to 18 years, with a Cobb angle between 10 and 25 degrees, will be included in the study. The subjects will be randomly divided into two groups; Schroth exercises will be applied to one group and pilates exercises will be applied to another group. All participants will participate in exercise sessions of 60 minutes a day, 3 days a week, for 8 weeks. Each participant will receive a total of 24 sessions of exercise therapy under the supervision of a physiotherapist. In this study, exercises that activate the muscle groups responsible for maintaining the correct posture and correcting the curvature will be selected for practice. Within the study, axial trunk rotation with a scoliometer, respiratory functions and respiratory muscle strength measurement with spirometry, functional capacity with the 6-minute walking test, balance with the Tecnobody balance measuring device, quality of life with Scoliosis will be assessed by the Research Society-22 Quality of Life Questionnaire. The results obtained from the study are of great importance as they will help to determine the effects of Schroth and pilates exercises on spinal deformity and the treatment of related problems in patients with AIS and to establish appropriate programs for the prevention and treatment of these problems.

ELIGIBILITY:
Inclusion Criteria:

* having a Cobb angle between 10 and 25 degrees
* age between 10-18 years

Exclusion Criteria:

* Presence of secondary scoliosis (congenital, muscular and neurological scoliosis)
* Presence of any cardiovascular and pulmonary disease that will prevent respiratory functions
* Having a history of thoracic surgery
* Use of assistive devices
* Presence of a secondary orthopedic problem

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
respiratory functions | 2 years
  These measurements include forced vital capacity (FVC), forced expiratory volume in one second (FEV1), and peak flow rate. (PEF), 25-75% flow rate of forced vital capacity (FEF25-75), expected values according to age, height, and weight and their percentages, and the ratio of forced expiratory volume in the first second to forced vital capacity (FEV1/FVC) will be recorded. MIP will be obtained by measuring the intraoral pressure during maximum inspiration against a closed valve for 1-3 seconds after maximum expiration. MEP will be obtained by measuring the intraoral pressure during maximum inspiration against a closed valve for 1-2 seconds after maximum inspiration.
spine structure | 2 years
  A scoliometer will be used to evaluate axial trunk rotation. Scoliometer is used to measure the rotational severity of the curvature of the vertebra in the horizontal plane. The patient will be asked to stand in a standing position, with the feet slightly open, stretching his arms forward and joining his hands with the palms facing each other. Then, he/she will be asked to lean forward until his/her body is horizontal by putting his/her hands between his/her knees without bending his/her knees. The scoliometer will be placed at the apex by the therapist positioned behind the patient, and the rotation value shown by the scoliometer will be recorded in degrees. While the interpersonal reliability of the scoliometer was found to be "excellent", its inter-measurement reliability was stated to be "very good".

SECONDARY OUTCOMES:
functional capacity | 2 years
  Functional capacity will be evaluated with the 6-minute walk test (6MWT), which is the most widely used because it is easily applicable. The test was performed according to the 6 WT criteria references determined by the American Thoracic Society. Individuals will be asked to walk as fast as possible without running in a 30-meter straight corridor for six minutes.
balance | 2 years
  Balance will be assessed with the Tecnobody Balance Measurement Device. Individuals step on the device, first of all, individuals will be informed about how the tests will be applied. A repeat test will be performed before each test to ensure adaptation and familiarization with the device. Individuals' postural sway and stability limits will be evaluated. In the postural sway evaluation, individuals will be asked to place their hands on their waist and maintain their balance, then to stand still with their eyes open for 30 seconds and then with their eyes closed for 30 seconds. In the stability limit evaluation, individuals will be asked to move the moving cursor to the square where the light is on and will be told not to lift their feet from the platform while doing this. The test will end after moving the cursor to the squares that light up in a total of eight different directions. Individuals will be given a 1-2 minute rest period between each test5.
quality of life of the participants | 2 years
  Participants' quality of life will be evaluated with SRS-22. SRS-22 is an easy and practical quality of life questionnaire designed specifically for scoliosis to evaluate the current condition of the spine.

CONTACTS AND LOCATIONS:
Overall Officials: sevtap gunay ucurum, Principal Investigator — İzmir Katip Çelebi University
Locations (2):
- Turkey (Türkiye) (2):
  - Izmir Katip Celebi University, Izmir
  - İzmir Katip Çelebi University, Izmir

IPD SHARING:
Plan to Share IPD: Undecided